CLINICAL TRIAL: NCT04005820
Title: Treatment for French Pediatric Patients With Renal Tumours According to the International SIOP Renal Tumour Study Group (RTSG) 2016 UMBRELLA Protocol Including Analysis of Tumour Chromosome 1q Gain and Central Radiology Review
Brief Title: Impact of Tumour 1q Gain in French Pediatric and Young Adult Patients With Renal Tumours
Acronym: UMBRELLA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-44
Record Dates: First submitted 2019-06-12; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Kidney Cancer
Keywords: pediatric
MeSH Terms: conditions — Kidney Neoplasms | interventions — Histocompatibility Testing; Tumor Burden; Urination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- children and young adults supported in one of SFCE's centers (Experimental)
  Interventions: Other: Radiologic Centralized Review; Other: Tissue sample (tumor, sung, urine)

INTERVENTIONS:
Other: Radiologic Centralized Review — The patient's imaging will be examined in one of the examination centers
Other: Tissue sample (tumor, sung, urine) — all the samples will be made during the patients care

SUMMARY:
French patients with nephroblastoma (Wilms tumour, WT) have been treated for > 40 years according to International Society of Paediatric Oncology (SIOP) protocols with currently 267 centres across 28 countries collaborating internationally within the SIOP Renal Tumour Study Group (RTSG).

Over the last decades more than 10,000 children have been prospectively enrolled in SIOP WT studies and trials. This has resulted in more standardised diagnostic procedures, improved risk stratification, and adjusted treatment recommendations for most renal tumours. The treatment of patients with renal tumours according to SIOP protocols include preoperative chemotherapy, surgery (tumour-nephrectomy + node-picking ± metastasectomy) followed by risk- and stage-based postoperative chemotherapy ± radiotherapy. Central pathology review is nowadays routinely performed in order to prevent misclassification of stage and histology risk group.

The current SIOP 2001 protocol has come to an end with as major achievement the scientific proof of omitting doxorubicin in stage II and III patients with as a consequence less risk of sequelae. Moreover, in the SIOP 2001 protocol, several tumour biological aspects have been assessed that seem to interfere with outcome (chromosomal gain of 1q, or loss of 1p and 16q, blastemal residual volume). Chromosomal 1q gain is considered to be present in 25-35% of patients with nephroblastoma with a negative impact on event-free survival (EFS) in retrospective analyses. These biological aspects will be studied prospectively as a primary objective in the new SIOP RTSG 2016 UMBRELLA protocol that integrates diagnostics, treatment and follow-up guidelines as well as several research projects.

The main mission of the International Society of Paediatric Oncology (SIOP) Renal Tumour Study Group (RTSG) is to increase survival and to reduce acute treatment toxicity and late effects in all children diagnosed with any renal tumour. In this context, SIOP RTSG is aiming to offer all these patients the same standardized high quality diagnostics and treatment, independent of the tumour type. The new SIOP RTSG 2016 integrated diagnostic and research UMBRELLA protocol serves as an entry for including all children with a renal tumour in the SIOP-RTSG centers, including prospective biomarker analyses. Subsequently, treatment is recommended according to the SIOP RTSG 2016 UMBRELLA treatment guidelines, which provides treatment strategies for all patients with Wilms tumour (WT) and other renal tumours. Central radiology review (CRR) has been proposed as a novel tool within the diagnostic UMBRELLA protocol in order to optimize the diagnostics and hence the treatment.

The definition of metastatic disease in WT remains difficult since pulmonary nodules may not always be of malignant origin. The differential diagnosis of a pulmonary lesion seen in a child with WT is broad. In addition to malignancy, it includes atelectasis, fibrosis, pneumonitis, subpleural lymph nodes, and other infectious or inflammatory lesions. In addition, the issue of "CT-only" nodules in WT and adequate treatment needs to be solved. In previous protocols, the treatment strategy was based on the diagnosis of pulmonary metastases (92% of all metastases) by conventional pulmonary X-ray. Patients with CT-only nodules (= nodules not visible on conventional X-ray) were supposed to be treated as having localized WT. However, retrospective analyses of SIOP series (Smets et al), showed that patients with CT-only nodules had a less favourable prognosis as compared to patients with truly localized disease with a 12% difference in three-year event-free survival.

The diagnostics of bilateral renal tumours (stage V) often is complicated since it may be difficult to distinguish true WT from nephroblastomatosis/ nephrogenic rests, a pre malignant renal (multifocal) anomaly, which may respond to preoperative chemotherapy. An optimal multi-disciplinary sequential diagnostic procedure is required in order to propose the best adapted therapeutic approach to preserve sufficient renal tissue.

ELIGIBILITY:
Inclusion Criteria:

* Children, adolescents or young adults (up to and including 30 years) with primary or relapsed renal tumor diagnosed at a participating SIOP-RTSG center
* Subject agreeing to participate

Exclusion Criteria:

* Absence of informed consent

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 510 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Impact of tumour chromosomal 1q gain on event-free survival (EFS) | 5 years
  5-year EFS will be analyzed by Kaplan-Meier analysis in all patients with nephroblastoma. The impact of tumour 1gain on 5-year EFS will be analyzed statistically by log-rank analysis comparing those patients with 1q gain with patients withour 1q gain
Impact of tumour chromosomal 1q gain on overall survival (OS) | 5 years
  5-year OS will be analyzed by Kaplan-Meier analysis in all patients with nephroblastoma. The impact of tumour 1gain on 5-year OS will be analyzed statistically by log-rank analysis comparing those patients with 1q gain with patients withour 1q gain

SECONDARY OUTCOMES:
Central radiology review | 5 years
  Central radiology review will be proposed as a novel tool in order to optimize the diagnostics and hence the treatment of patients with renal tumours. As such it will impact the 5-year EFS and OS.
Blastemal residual volume | 5 years
  The impact of balstemal residual volume > 10 ml in the tumour on outcome will be compared to patients with < 10 ml of residual volume. It is anticipated that ther ewill be a statisticla difference in EFS and/or OS.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — AP HM
Locations (1):
- Service d'Hématologie-Oncologie Pédiatrique - APHM, Marseille, France